CLINICAL TRIAL: NCT05453721
Title: Effect and Long-Term Outcomes of Indocyanine Green Fluorescence Imaging Method Versus Modified Inflation-Deflation Method in Identification of Intersegmental Plane: A Multicenter、Prospective、Randomized Controlled Trial
Brief Title: Effect and Long-Term Outcomes of Indocyanine Green Fluorescence Imaging Method Versus Modified Inflation-Deflation Method in Identification of Intersegmental Plane（IMPLANE-0529）
Acronym: IMPLANE-0529
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Nanchang University (Other)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Dazhou Central Hospital (Other); Ningde Municipal Hospital of Ningde Normal University (Unknown); First Affiliated Hospital of Gannan Medical University (Other); Fuzhou Pulmonary Hospital of Fujian (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Ningbo No.2 Hospital (Other); Guangdong Provincial People's Hospital (Other); Zhejiang Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Jian Tang, M.D., Ph.D, Professor, The First Affiliated Hospital of Nanchang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFTS-1
Record Dates: First submitted 2022-06-24; First posted 2022-07-12 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Segmentectomy; Non-small Cell Lung Cancer Stage I
Keywords: Segmentectomy; Intersegmental plane identification; Indocyanine green fluorescence imaging method; Modified inflation-deflation method
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: This study has two parallel arms, Indocyanine green fluorescence imaging method (treatment arm) and Modified inflation-deflation method (control arm) are included in this study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Indocyanine green fluorescence imaging method group (Experimental): Using indocyanine green fluorescence imaging method to identify intersegmental plane in segmentectomy
  Interventions: Procedure: Indocyanine green fluorescence imaging method
- Modified inflation-deflation method group (Active Comparator): Using modified inflation-deflation method to identify intersegmental plane in segmentectomy
  Interventions: Procedure: Modified inflation-deflation method

INTERVENTIONS:
Procedure: Indocyanine green fluorescence imaging method — Using indocyanine green fluorescence imaging method to identify intersegmental plane in segmentectomy
  Arms: Indocyanine green fluorescence imaging method group
Procedure: Modified inflation-deflation method — Using modified inflation-deflation method to identify intersegmental plane in segmentectomy
  Arms: Modified inflation-deflation method group

SUMMARY:
This study is a multi-center, prospective, randomized controlled clinical trial. The purpose is to compare the difference of indocyanine green fluorescence imaging method and modified inflation-deflation method in identifying intersegmental plane in segmentectomy, and provide high-level evidence for the selection of intersegmental plane identification method in early NSCLC segmental resection.

DETAILED DESCRIPTION:
In patients with early-stage lung cancer, segmentectomy has comparable long-term survival results compared with conventional lobectomy, but patients have a higher postoperative quality of life because more lung tissue is preserved.

Segmentectomy is based on accurate anatomy, and the identification of intersegmental plane is one of the keys to accurate anatomy of segmentectomy.

At present, differential ventilation and differential colorimetry are clinically used to cause the difference between the target segment and the adjacent lung segment to identify intersegmental plane, which both have advantages and disadvantages. Clinical consensus on the best method for intersegmental plane identification has not been formed.

This study is a multi-center, prospective, randomized controlled clinical trial. The study plans to enroll 272 patients with peripheral stage I NSCLC with tumor diameter ≤2cm and consolidation tumor rate <1. Eligible patients will be randomly divided into the experimental group (indocyanine green fluorescence imaging method) or control group (modified inflation-deflation method) at a ratio of 1:1.

This study is expected to compare the difference of indocyanine green fluorescence imaging method and modified inflation-deflation method in identifying intersegmental plane in segmentectomy, and provide high-level evidence for the selection of intersegmental plane identification method in early NSCLC segmentectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 80 years old;
2. According to the surgical standards of the Eighth edition of People's Medical Publishing House, patients whose blood pressure was under 160/100mmHg and blood glucose was under 5.6-11.2mmol /L with normal functions of major organs such as heart, lung, liver and kidney before surgery are included. The main criteria are as follows:

   i. Cardiac function examination indicated Goldman index grade 1-2; ii. Pulmonary function examination suggested postoperative predicted FEV1≥40% and DLCO≥40%; iii. Total bilirubin ≤1.5 times the upper limit of normal; iv. Alanine aminotransferase and aspartate aminotransferase ≤2.5 times the upper limit of normal value; v. Creatinine ≤1.25 times the upper limit of normal value and creatinine clearance ≥60ml/min;
3. The center of the lesion is located in the other lobes except the middle lobe, and in the middle and outer third of the lung;
4. The maximum diameter of the tumor was not more than 2cm on TLC(Thin layer CT) scan and the clinical stage was cT1a-1bN0M0(according to AJCC staging criteria, eighth edition);
5. Consolidation tumor rate <1；
6. ECOG PSscore 0-1;
7. All relevant examinations should be completed within 28 days before surgery;
8. Patients who understand the study and have signed informed consent.

Exclusion Criteria:

1. Patient with a history of iodine or indocyanine green allergy;
2. Patient who had received antitumor therapy (radiotherapy, chemotherapy, targeted therapy, immunotherapy) prior to surgery;
3. Patient with a history of other malignancies;
4. Patient with secondary primary cancer at enrollment;
5. Small cell lung cancer;
6. Prior history of unilateral thoracotomy;
7. Woman in pregnant or breastfeeding period;
8. Patient with interstitial pneumonia, pulmonary fibrosis or severe emphysema;
9. An active bacterial or fungal infection that is difficult to control;
10. Severe mental illness;
11. History of severe heart disease , heart failure , myocardial infarction or angina pectoris within the last 6 months;
12. patient that researcher considers inappropriate to participate in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2022-08-04 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Success rate of intersegmental plane identification | During the operation
  Successful intraoperative appearance of the intersegmental plane is considered a success

SECONDARY OUTCOMES:
Intersegment plane identification time | During the surgery
  Indocyanine green injection/start of ventilation to the first observed intersegment plane appearance
Surgery time | During the surgery
  Time from the beginning to the end of the surgery
Intraoperatve blood loss | During the surgery
  Blood loss during the surgery
Postoperative blood loss | Postoperative in-hospital stay up to 30 days
  Blood loss after the surgery
Postoperative air leakage rate | Postoperative in-hospital stay up to 30 days
  Air leakage after the surgery
Postoperative air leakage time | Postoperative in-hospital stay up to 30 days
  time of air leakage after the surgery
Preoperative pulmonary function | 1 week before the surgery
  FEV1.0(forced expiratory volume in 1.0 s)
Preoperative pulmonary function | 1 week before the surgery
  FVC(forced vital capacity)
Postoperative pulmonary function | 6/12 months after surgery
  FEV1.0(forced expiratory volume in 1.0 s)
Postoperative pulmonary function | 6/12 months after surgery
  FVC(forced vital capacity)
Quality of life（EORTCQLQ-C30) | 6/12 months after surgery
  Quality of life Scale
Adverse event rate | Through study completion, an average of 2 year
  According to CTCAE-V5.0
Adverse event level | Through study completion, an average of 2 year
  According to CTCAE-V5.0
Surgical complication | Postoperative in-hospital stay up to 30 days
  According to Clavien-Dindo grading system
Postoperative 30-day mortality | Within 30 days after surgery
  Deaths occurring within 30 days after surgery
Postoperative 90-day mortality | Within 90 days after surgery
  Deaths occurring within 90 days after surgery
Reoperation rate | Within 30 days after surgery
  The percentage of patients who need a second operation
Number of stapler nail bin used for cutting | During the surgery
  Number of stapler nail bin used for cutting
R0 resection rate | Within 14 days after surgery
  Negative surgical margin under the microscope

OTHER OUTCOMES:
Coincidence rate of intersegmental plane identification | Within 14 days after surgery
  The shortest distance between the nodule and the cutting edge in all directions in postoperative pathological specimens versus distances measured in preoperative 3D reconstruction in same directions

CONTACTS AND LOCATIONS:
Overall Officials: Jian Tang, M.D., Ph.D, Principal Investigator — The First Affiliated Hospital of Nanchang University
Locations (1):
- The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No